CLINICAL TRIAL: NCT02861053
Title: Inflammatory Bowel Disease : Could a Regular Physical Activity Reduce Patients Fatigue ?
Acronym: MICI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016/013/HP
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chronic quiet inflammatory bowel disease patient (IBD) (Experimental): Patient with chronic quiet inflammatory bowel disease patient (IBD) with regular and moderate physical activity
  Interventions: Other: regular and moderate physical activity; Other: No regular and moderate physical activity more than usual
- chronic quiet inflammatory bowel disease Patient (IBD) (Sham Comparator): Patient with chronic quiet inflammatory bowel disease patient (IBD) with no regular and moderate physical activity more than usual
  Interventions: Other: regular and moderate physical activity; Other: No regular and moderate physical activity more than usual

INTERVENTIONS:
Other: regular and moderate physical activity — regular and moderate physical activity will be done 3 times per week more than usual
Other: No regular and moderate physical activity more than usual — regular and moderate physical activity will be done as usual

SUMMARY:
The chronic fatigue is observed in approximately 40 % of the patients with a chronic quiet inflammatory bowel disease (IBD) and impacts the quality of life of the patients. The beneficial role of a regular physical activity on the quality of life of patients having an IBD was demonstrated in 5 studies including only 1 controlled one [Bilski, on 2013]. The mechanism by which the physical activity could improve the quality of life of the patients remains unknown (stress decreased, reduction of the inflammatory process) [Bilski, on 2014]. Several studies concerning other chronic pathologies such as fibromyalgia, have demonstrated the beneficial effect of a regular physical exercise to reduce the fatigue of patients. It was recently demonstrated that the chronic fatigue observed in patients with IBD came along with a physical reduction in the performances during the exercise test and a reduction in the physical activity of the patients [Vogelaar, 2015].

Our hypothesis is that a regular moderate physical activity could improve physical performance during an effort et could reduce the chronic fatigue and improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Patients suffering from IBD
* Patients with a FACIT score < 30
* Patients with BD in remission with a C-reactiv protein dose < 5
* Patients with Hemoglobin dosage > 10g/dl
* Patients with 18<BMI<30 kg/m2
* Informed consent given by the patients
* Patients affiliated to the social security
* Patients living not far from the centre where the rehabilitation program will be performed
* Women with no risk of pregnancy (menopausal women or with contraceptive drugs).

Exclusion Criteria:

* Patients ≥ 45 years old
* Inability to walk or to ride a bike
* Contraindication to practice physical exercise
* Contraindication to exercise test
* Participation to another research study within the week preceding the beginning of the protocol
* Patients unstable smokers
* Patients unable to keep their medical treatment stable along the study
* Patients with a regular intensive physical practice
* Patients with depression (HAD>11/21)
* Patients with bad sleep quality (PSQI score >5)
* Pregnant or breast-feeding patients
* Patients under legal protection

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Difference from baseline in the evaluation of fatigue | 3 Month
  Evaluation of fatigue using FACIT questionnaire

SECONDARY OUTCOMES:
Difference from baseline in the Evaluation of the Quality of life | 3 Month
  Evaluation of the Quality of life using Quality of life scores (IBDQ)
Difference from baseline in the Evaluation of the Quality of life | 3 Month
  Evaluation of the Quality of life using Quality of life scores (SF36)

CONTACTS AND LOCATIONS:
Overall Officials: David DEBEAUMONT, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: Undecided